CLINICAL TRIAL: NCT07295782
Title: Fibrin Clot Properties and Thrombin Generation in Women After Urogynecological Surgery.
Brief Title: The Assessment of Fibrin Clot Phenotype and Thrombin Generation in Women After Urogynecological Surgeries.
Status: Recruiting | Type: Observational
Sponsor: Jagiellonian University (Other)
Responsible Party: Principal Investigator, Magdalena Piróg, MD, MD, PhD, Jagiellonian University
Other Study IDs: 1072.6120.315.2022
Record Dates: First submitted 2025-12-08; First posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Uterine Prolapse; Urine Incontinence
Keywords: uterine prolapse; urine incontinence; fibrin clot; fibrinolysis; thrombin
MeSH Terms: conditions — Uterine Prolapse; Nocturnal Enuresis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women with urine incontinence/ uterine prolapse: Healthy women with urine incontinence/ uterine prolapse qualified for urogynecological surgery
  Interventions: Diagnostic Test: determination of fibrin clot properties

INTERVENTIONS:
Diagnostic Test: determination of fibrin clot properties — Determination of fibre clot properties and thrombin generation in women with uterine prolapse/ urine incontinence before and after urogynecological surgery.

SUMMARY:
Determination of fibrin clot properties along with thrombin generation in women after urigynecological surgery.

DETAILED DESCRIPTION:
Fibrin clot permeability and susceptibility to lysis along with thrombin generation

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70
* treatment failure (pharmacotherapy) due to uterine prolapse or urine incontinence

Exclusion Criteria:

* prolonged thromboprophylaxis
* planned surgery other than due to urine incontinence/uterine prolapse
* acquired or congenital thrombophilia

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Participants with urine incontinence and uterine prolapse will be enrolled.
Study Population: Women with diagnosed uterine prolapse or urine incontinence after failure of pharmacotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-12-10 (Estimated); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
fibrin clot phenotype | December 2025 till May 2026
  fibrin clot permeability and susceptibility to lysis
Thrombin generation | December 2025 till May 2026
  Endogenous thrombin generation

CONTACTS AND LOCATIONS:
Locations (1):
- Gynecological Endocrinology Department, Krakow, Małopolska, Poland